CLINICAL TRIAL: NCT05679089
Title: Assessment of Early Detection Based on Liquid Biopsy in Intracranial Tumors: a Prospective Observational Study
Brief Title: AssesSment of Early deteCtion basEd oN liquiD Biopsy in Intracranial Tumors
Acronym: ASCEND-BRAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2022009
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Tumors
Keywords: intracranial tumors, early detection, liquid biopsy, cell-free DNA methylation
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer Arm: Participants with newly diagnosed intracranial malignant tumors, from whom blood samples will be collected.
  Interventions: Device: early detection test
- Benign Arm: Participants with newly diagnosed benign central nervous system disorders, from whom blood samples will be collected.
  Interventions: Device: early detection test
- Healthy arm: Participants without known presence of malignancies or certain benign diseases, from whom blood samples will be collected.
  Interventions: Device: early detection test

INTERVENTIONS:
Device: early detection test — Blood collection and early detection testing

SUMMARY:
ASCEND-BRAIN is a prospective, observational study aimed at early-detection of intracranial tumors by combined assays of cfDNA methylation and other biomarkers. The study will enroll approximately 358 participants including intracranial malignant tumors, patients with benign disorders of central nervous system and healthy participants.

ELIGIBILITY:
Inclusion Criteria for Cancer Participants:

* Age 40-75 years
* Ability to provide a written informed consent
* Pathologically confirmed diagnosis or highly suspicious cases of intracranial malignant tumors
* No prior or ongoing anti-cancer treatment (local or systematic) prior to study blood draw

Inclusion Criteria for Benign Disease Participants:

* Age 40-75 years
* Ability to provide a written informed consent
* Pathologically confirmed diagnosis or highly suspicious cases with benign disorders of central nervous system
* No prior or ongoing radical treatment of the benign disorders of central nervous system prior to study blood draw

Inclusion Criteria for Healthy Participants

* Age 40-75 years
* Ability to provide a written informed consent
* No cancer-related symptoms or other uncomfortable symptoms prior to study blood draw

Exclusion Criteria for All Participants:

* Insufficient qualified blood samples
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
* Recipient of blood transfusion within 7 days prior to blood draw
* Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw, such as rheumatic drugs (methotrexate, cyclophosphamide, or azathioprine), or endocrine drugs (tamoxifen)

Additional Exclusion Criteria for Cancer Participants:

-Other current malignant diseases or multiple primary tumors

Additional Exclusion Criteria for Benign Disease Participants:

-Current or history of malignancies

Additional Exclusion Criteria for Healthy Participants:

* Recipient of anti-infectious therapy within 14 days prior to study blood draw
* Prior or ongoing treatment of cancer within 3 years prior to study blood draw
* Current autoimmune disease or clinically significant or uncontrolled comorbidities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the participating medical center and assigned into three arms, including participants with newly diagnosed intracranial malignant tumors, benign disorders of central nervous system and healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of a cfDNA methylation-based early detection model for intracranial tumors. | 12 months

SECONDARY OUTCOMES:
The sensitivity and specificity of a cfDNA methylation-based early detection model for intracranial tumors of different grades(WHO I-IV) and mutant subtypes(IDH mutant/wild type). | 12 months

OTHER OUTCOMES:
The specific cfDNA methylation landscape of intracranial tumors in China | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Guo, MD,Ph.D, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China